CLINICAL TRIAL: NCT05146986
Title: Prospective Multi-center Comparative Study of RibFix Blu Thoracic Fixation System Versus Non-surgical Treatment in Non-flail Chest Rib Fractures
Brief Title: RibFix Blu Thoracic Fixation System Versus Non-surgical Treatment in Non-flail Chest Rib Fractures
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSA2021-16SU
Record Dates: First submitted 2021-10-15; First posted 2021-12-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Rib; Fracture
Keywords: Non-flail chest
MeSH Terms: conditions — Rib Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Non-surgical group: Patients will receive analgesia and symptomatic management treatment
  Interventions: Device: Non surgical and Surgical
- Surgical group: Patients will receive surgical treatment using RibFix Blu Thoracic Fixation System
  Interventions: Device: Non surgical and Surgical

INTERVENTIONS:
Device: Non surgical and Surgical — For non-surgical group, patients will receive non-surgical treatment (analgesia and symptomatic management treatment).
  For surgical group, patients will receive surgical treatment using RibFix Blu Thoracic Fixation System.

SUMMARY:
This is a prospective, multi-center, observational, cohort study involving skilled cardiothoracic surgeons who are experienced in implanting the treatment of non-flail chest rib fractures and the use of RibFix Blu Thoracic Fixation System.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the benefits of surgical stabilization of rib fractures (SSRF) in patients with non-flail chest rib fractures using RibFix Blu Thoracic Fixation System when compared to non-surgical (analgesia and symptomatic management) treatment. The study will include up to 167 cases of non-flail chest rib fractures with 95 cases in non-surgical treatment group and 72 cases in the surgical group. Each center may enroll up to maximum 30 cases to permit the assessment of outcome across a variety investigators and clinical settings. Enrolment will be competitive among sites and closed as soon as a total of 167 cases are recruited.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above (inclusive)
* Simple rib fracture with ≥ 3 consecutive ribs, and the broken ends showed clear displacements
* Indicated for surgical repair of rib fractures using RibFix Blu Thoracic Fixation System or non-surgical treatment (analgesia and symptomatic management treatment)
* Willing and able to complete scheduled follow-up evaluations as described in the study protocol
* Has participated in the Informed Consent process and is willing and able to sign an Institutional Review Board or Ethics Committee (IRB/EC) approved Patient Information/ Informed consent Form (PICF)

Exclusion Criteria:

* Flail chest rib fractures based on radiological or clinical findings
* Previous rib fractures or pulmonary problems, requiring continuous oxygen use at home pre-trauma
* Presence of any serious medical issues that placed patient in generally poor conditions such that he or she could not tolerate the surgery
* Chest trauma associated with severe craniocerebral injury, abdominal organ injury, severe spinal injury, limb fracture, or pelvic fracture requiring long-term bed rest
* Has serious medical disease that is a contraindication for general anesthesia, such as cerebral infarction, myocardial infarction and hemorrhagic syndrome
* Any contraindications listed in the manufacturer's Instruction to use for RibFix Blu Thoracic Fixation System as per below:

  * Spanning a midline sternotomy
  * Active Infection
  * Foreign body sensitivity
* Is known to be pregnant
* Is a prisoner, known alcohol or drug user or mentally incompetent or unable to understand what participation in this study entails.
* Participation in another surgical intervention that may influence any of the outcome parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-flail chest rib fractures who plan to receive surgical treatment with RibFix Blu Thoracic Fixation System or non-surgical treatment, and meet the inclusion criteria and do not meet any exclusion criteria will be eligible to participate in the study
Sampling Method: Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Thoracic pain as assessed by numeric Rating Scale (NRS) | 2 weeks
  Level of thoracic pain determined using a numeric Rating Scale (NRS). Thoracic pain will be determined using an 11-point Numeric Rating Scale (NRS) in which 0 implicates no pain and 10 the worst pain. If a subject is not able to provide a response to the level of thoracic pain,

SECONDARY OUTCOMES:
Rate of Analgesic use | 12 weeks
  Analgesic use by the difference groups
Length of Hospital stay | 12 weeks
  Length of Hospital stay by the difference groups
Quality of life using EuroQoL-5L | 2 weeks, 6 weeks and 12 weeks
  Health related qualify of life using EuroQoL-5L(EQ-5D-5L) questionnaires from the different groups.
  A standardized measure of health-related quality of life states consisting of 5 dimensions, namely mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L version was used in the study. Each dimension has 5 responses recording 5 levels of severity (no problems/slight problems/moderate problems/severe problems or extreme problems). The responses to the EQ-5D dimensions are used to obtain a single EQ-5D index value where 1 represents full health and 0 represents death. The questionnaire also includes a vertical, visual analogue scale (EQ VAS) for the respondents to record their self-rated health where the 2 extreme ends of the scale are labelled as 'Best imaginable health state' and 'Worst imaginable health state' respectively
Pulmonary function | 12 weeks
  Pulmonary function will be assessed by the measuring the forced vital capacity (FVC) using a spirometer.
Pulmonary function | 2 weeks, 6 weeks and 12 weeks
  Pulmonary function will be assessed by the measuring the forced expiratory volume (FEV) using a spirometer.
Number of Participants with respiratory complications | 2 weeks, 6 weeks and 12 weeks
  Complications from the different groups assessed to be related to respiratory.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Marasco, Professor, Principal Investigator — The Alfred
Locations (5):
- Australia (3):
  - Hunter New England Health District, Sydney, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Alfred (Alfred Health), Melbourne, Victoria
- South Korea (2):
  - Yonsei Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Ajou University Hospital, Suwon, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: No